CLINICAL TRIAL: NCT03083067
Title: A Prospective Study of Salvational Intervention With ICS/LABA for Reducing Chronic Obstructive Pulmonary Disease Exacerbation Under Severe Air Pollution (SIRCAP) in Beijing
Brief Title: Salvational Intervention for Reducing AECOPD Under Severe Air Pollution
Acronym: SIRCAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University First Hospital (Other)
Collaborators: Peking University Shougang Hospital (Other); People's Hospital of Beijing Daxing District (Other); Beijing Jingmei Group General Hospital (Unknown); Beijing Miyun Hospital (Unknown); The Hospital of Shunyi District Beijing (Unknown); Beijing Luhe Hospital (Other); Civil Aviation General Hospital (Other); Beijing Jishuitan Hospital (Other); Aerospace 731 Hospital (Other); Beijing Changping Hospital (Unknown)
Responsible Party: Principal Investigator, Guangfa Wang, Prof. & MD., Peking University First Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SF2016-1-4071
Record Dates: First submitted 2017-03-03; First posted 2017-03-17 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: COPD Exacerbation; Air Pollution
Keywords: AECOPD; air pollution; COPD; salvational Intervention
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Budesonide, Formoterol Fumarate Drug Combination; Tiotropium Bromide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Salvational intervention(SI) group (Experimental): Budesonide/formoterol（160ug/4.5ug）will be used as an intervention drug on the foundation of original treatment.
  Interventions: Drug: Budesonide/formoterol; Drug: tiotropium bromide
- Control(CT) group (Active Comparator): CT group maintain the original treatment
  Interventions: Drug: tiotropium bromide

INTERVENTIONS:
Drug: Budesonide/formoterol — On the foundation of basic treatment strategies, inhaled budesonide/formoterol（160ug/4.5ug）will be used as an intervention drug for patients in PIC group. When air quality index (AQI) is above 200, they will temporary add one inhalation of budesonide/formoterol（160ug/4.5ug）twice a day until the third day after AQI drops below 200.
  Arms: Salvational intervention(SI) group
Drug: tiotropium bromide — Inhaled tiotropium bromide(18ug) will be used as routine medicine according to doctor's advice.

SUMMARY:
This is a multi-center, prospective, randomized and standard treatment parallel control clinical trial.A total of 764 stable COPD patients according to GOLD will be recruited and equally divided into two parallel groups, salvational intervention group (SI group) and control group (CT group).On the foundation of basic medicine, inhaled ICS/LABA will be used as an intervention drug for patients in SI group on severe air pollution days. It is aimed to evaluate whether this novel treatment strategy will decrease the frequency of AECOPD per year.

DETAILED DESCRIPTION:
This is a multi-center, prospective, randomized and standard treatment parallel control clinical trial. A total of 764 stable COPD patients with history of exacerbation according to GOLD will be recruited and equally divided into two parallel groups, salvational intervention group (SI group) and control group (CT group). The randomization is stratified by medical center and the random code is designed in a 1:1 ratio. The Department of Respiratory and Critical Care of Peking University First Hospital is responsible for this research. Other 10 units participating in the study include Peking University Shougang Hospital, People's Hospital of Beijing Daxing District, Beijing Jingmei Group General Hospital, Beijing Miyun Hospital, Beijing Changping Hospital, The Hospital of Shunyi District Beijing, Beijing Luhe Hospital Capital Medical University, Civil Aciation General Hospital, Beijing Jishuitan Hospital and Aerospace 731 Hospital. These 11 centers approximately cover area from urban to suburbs in Beijing.

Inhaled tiotropium bromide(18ug), budesonide/formoterol（160ug/4.5ug）or tiotropium bromide(18ug)+ budesonide/formoterol （160ug/4.5ug）will be used as basic medicine. On the foundation of basic medicine, inhaled budesonide/formoterol（160ug/4.5ug）will be used as an intervention drug for patients in SI group. When air quality index (AQI) is above 200, they will temporary add one inhalation of budesonide/formoterol（160ug/4.5ug）twice a day until the third day after AQI drops below 200. CT group maintains the original treatment. Besides baseline, patients will be formally visited 4 or 5 times during this trial: before randomization (for those who need pharmacological washout) and every six months after randomization.

Primary outcome is the frequency of AECOPD per year, which is defined as the frequency of AECOPD/the number of patients/year. Secondary outcomes include the number of unplanned outpatient visits, emergency medical visits, hospitalization, medical expense and mortality caused by AECOPD per year.

The study protocol has been approved by the Peking University First Hospital Institutional Review Board (IRB) (2016[1032]). Any protocol modifications will be submitted for the IRB review and approval.

ELIGIBILITY:
Inclusion Criteria:

1. aged at 40-80 years old;
2. spirometry confirmed diagnose of COPD with at least once exacerbation before, and stable for at least three months;
3. quit smoking for more than six months;
4. be able to engage in daily activities;
5. have willing to participate in this study, follow the research program and have the ability to sign the informed consent;
6. Beijing residents;
7. can be contacted;

Exclusion Criteria:

1. history of asthma, lung cancer, active pulmonary tuberculosis, bronchiectasis, diffuse lung disease (interstitial pneumonia, pulmonary sarcoidosis, occupational lung disease, sarcoidosis et al) and pleural disease;
2. history of lobectomy and / or lung transplantation;
3. predicted life expectancy less than 3 years;
4. history of severe psychiatric illnesses, mental disorders, neurological disorders, malignant tumors, chronic liver disease, heart failure, autoimmune diseases, chronic kidney disease;
5. Never engage in outdoor activities;
6. plan to move out of Beijing in 3 years
7. Plan to carry out an indoor redecoration during the study;
8. Alcoholism, drug abuse or abuse of toxic solvents;
9. Allergic to the study drug or its ingredients, or have a clear contraindication of it;
10. Participation in another clinical trial;
11. Cannot finish long term follow-up or poor compliance;
12. Do not provide consent.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 402 (Actual)
Dates: Start 2017-03-20 (Actual); Primary Completion 2022-03-16 (Actual); Study Completion 2022-03-16 (Actual)

PRIMARY OUTCOMES:
the frequency of exacerbation of COPD per year | 3 year

SECONDARY OUTCOMES:
the number of unplanned outpatient visits caused by exacerbation of COPD per year | 3 years
the number of unplanned emergency medical visits caused by exacerbation of COPD per year | 3 years
the number of unplanned hospitalization caused by exacerbation of COPD per year | 3 years
the cost of unplanned medical expense caused by exacerbation of COPD per year | 3 years
the number of unplanned mortality caused by exacerbation of COPD per year | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Guangfa Wang, MD, Study Chair — Peking University First Hospital
Locations (11):
- China (11):
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Aerospace 731 Hospital, Beijing, Beijing Municipality
  - Beijing Changping Hospital, Beijing, Beijing Municipality
  - Beijing Jingmei Group General Hospital, Beijing, Beijing Municipality
  - Beijing Jishuitan Hospital, Beijing, Beijing Municipality
  - Beijing Luhe Hospital, Beijing, Beijing Municipality
  - Beijing Miyun Hospital, Beijing, Beijing Municipality
  - Civil Aviation General Hospital, Beijing, Beijing Municipality
  - Peking University Shougang Hospital, Beijing, Beijing Municipality
  - People's Hospital of Beijing Daxing District, Beijing, Beijing Municipality
  - The Hospital of Shunyi District Beijing, Beijing, Beijing Municipality

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhou T, Zhong Y, Liao J, Wang G, Li X, Qian X, Xiang P, Chen X, Xu Z, Zhang F, Wang X, Wang S, Li X, Yu C, Zhang Y, Xia G, Dai L. A prospective study of salvational intervention with ICS/LABA for reducing chronic obstructive pulmonary disease exacerbation under severe air pollution (SIRCAP) in Beijing: protocol of a multi-center randomized controlled trial. BMC Pulm Med. 2019 Jan 25;19(1):22. doi: 10.1186/s12890-018-0771-9. PMID 30683080